CLINICAL TRIAL: NCT01981265
Title: Genome-wide Study for Disease Susceptibility Gene(s) in Patients With Hand Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201109024RC
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Hand Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hand osteoarthritis

SUMMARY:
This is a case-control study involving one medical center and one research institute to develop a data-set containing a minimum of 100 osteoarthritis cases, minimum of 100 independent controls of similar gender ratio and a minimum of 100 disease controls (cases with hip and/or knee OA) to associate DNA sequence (allelic) variations in candidate genes with osteoarthritis phenotypes.

This study is intended to begin at the Institute of Biomedical Sciences at Academia Sinica (which includes National Genotyping Center (NGC) and National Clinical Core (NCC)), National Taiwan University Hospital.

ELIGIBILITY:
Exclusion Criteria:

1. Patients with the following diseases will be excluded：Rheumatoid arthritis, Gout arthritis, Psoriatic arthropathy, Hypertrophic osteoarthropathy, Hypermotility syndrome, Hemochromatosis, Post-traumatic OA, Other secondary-form OA and Lupus.
2. The individual is excluded if the hand X-rays show MCP changes compatible with hemochromatosis. The site then is obligated to measure fasting transferrin saturation (FE/TIBC ratio) and if >55%, the individual is excluded.
3. Have more than 3 swollen MCP joints equal to, or greater than KL grade 2.
4. Be unable to give informed consent.
5. One cannot participate in this study if other members of his or her immediate family have already been recruited (Only one person from each family can participate in the study).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Participating patients must be at least 45 years of age.
  2. All Patients must have radiographic hand OA.
  3. All Patients must be of Han Chinese ethnic background.
  4. Enrolled participants must give voluntary written consents to participate in this study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Hand Osteoarthritis related gene expression assay | 4 years
  The sample was collected from the patient who suffered from osteoarthritis of finger joints, espcially DIP joint. The operation was perfomed due to arthrodesis procedure. So we set the outcome measurement goal for the arthrodesis successful rate.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hao Chang, Study Director — Department of Orthopedics, National Taiwan University Hospital and National Taiwan University College of Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan